CLINICAL TRIAL: NCT01462383
Title: The Role of the EKG in Anticancer Phase I Drug Development
Brief Title: The Role of the EKG in Anticancer Drug Development
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: DR11-0061
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Malignancy; Cardiac complications; Electrocardiograms; ECG; Chart Review; Data Review; Data Analysis; Phase I; Clinical Research Study
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Primary Objective:

-Evaluate incidence of cardiac complications in Phase I patients.

Secondary Objective:

-To identify variables (i.e. number of electrocardiograms (EKG) performed) that lead to the detection of cardiac events.

DETAILED DESCRIPTION:
The research plan includes a retrospective review of the chart of past UT MD Anderson Cancer Center (MDACC) patients and the experience in treating them.

All studies analyzed will be Phase I clinical trials.

Analysis is designed to collect information on the number of and timeframe within which ECGs are performed on these trials. Data on adverse events and serious adverse events, dose modifications based on ECG changes, attribution to drug, incidence and types of ECG changes specifically QTC prolongation as well as their influence on study procedures like dose limiting toxicities (DLTs) in dose escalation phase of the studies.

Study conducted using clinical records of patients treated on Phase I protocols in the MDACC Department of Investigational Cancer Therapeutics. The demographic data to be collected from patients whose charts will be analyzed will include variables such as age, gender, primary cancer, stage of the disease, performance status, treatment characteristics (i.e., number and type of prior therapies), disease status, adverse events, laboratory data (i.e., complete blood count/differential/platelets, tumor markers), and treatment outcomes.

The analysis will allow identification and descriptive analysis of the occurrence of cardiac events in the phase I population and will help define the role of protocol required EKGs in their detection.

HIPAA privacy and confidentiality guidelines will be followed. The database will be secured in the Department server. A Data coordinator has been recruited to undertake this project. The information derived from these observations will help the investigators formulate research questions and projects to develop future prospective studies.

The statistical analysis will be performed in a descriptive fashion with paired and multivariable analyses.

The analyses will be reported using summary tables, figures, and data listings. Continuous variables will be summarized using the mean, standard deviation, median, minimum, and maximum.

This study will be conducted at the MD Anderson Cancer Center in Houston, Texas.

ELIGIBILITY:
Inclusion Criteria:

* All types of advanced cancer

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients in the Department of Investigational Cancer Therapeutics diagnosed with a malignancy and registered at MDACC for medical care on IRB approved sponsored protocols active between January 1, 2006 and December 31, 2009.
Sampling Method: Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Cardiac Complications in Participants on Phase I Protocols | 3 years
  Data review of studies, active between January 1, 2006 and December 31, 2009, who included ECGs in their safety evaluations. Use of identification and descriptive analysis of cardiac events occurrence in the phase I population to define role of protocol required EKGs in their detection. Statistical analysis performed in a descriptive fashion with paired and multivariable analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.utmdanderson.org